CLINICAL TRIAL: NCT03428412
Title: Effects of Traditional Chinese Medicine on AECOPD Patients: A Multi-center, Randomized, Double-blind, Controlled Trial
Brief Title: Effects of Traditional Chinese Medicine on AECOPD Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for AECOPD
Record Dates: First submitted 2018-01-19; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Acute Exacerbation; Medicine, Chinese Traditional
Keywords: Chronic Obstructive Pulmonary Disease; Acute exacerbation; Traditional Chinese medicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM plus conventional drug (Experimental): The experimental group will receive three type of TCM in addition conventional drug according to 2017 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines for AECOPD.
  Interventions: Drug: TCM and conventional drug
- TCM placebo plus conventional drug (Placebo Comparator): The control group will receive three type of placebo TCM in addition conventional drug according to 2017 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines for AECOPD.
  Interventions: Drug: TCM placebo and conventional drug

INTERVENTIONS:
Drug: TCM and conventional drug — All patients were treated with medicine based on 2017 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines for AECOPD.
  The Experimental group will receive TCM according to the TCM syndrome. Sanhanhuayin granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of external cold and internal fluid in 14 treatment days.
  Qingrehuatan granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of phlegm-heat congesting lung in 14 treatment days.
  Zaoshihuatan granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of phlegm-damp amassing in lung in 14 treatment days.
  Arms: TCM plus conventional drug
Drug: TCM placebo and conventional drug — All patients were treated with medicine based on 2017 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines for AECOPD.
  The control group will receive TCM placebo according to the TCM syndrome. Placebo Sanhanhuayin granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of external cold and internal fluid in 14 treatment days.
  Placebo Qingrehuatan granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of phlegm-heat congesting lung in 14 treatment days.
  Placebo Zaoshihuatan granule (Jiangyin Tian Jiang Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for syndrome of phlegm-damp amassing in lung in 14 treatment days.
  Arms: TCM placebo plus conventional drug

SUMMARY:
This is a multi-center, randomized, double-blind, controlled trial to compare the efficacy of two therapies for patients with AECOPD. 378 subjects will be randomly assigned to one therapies (conventional drug, and the combination of conventional drug and TCM) for 14 days treatment. After the treatment period, subjects in two arms will be followed up for 4 weeks. The primary outcomes will include COPD Assessment Test (CAT), and secondary outcomes include treatment failure rate, treatment success rate, hospitalization time, hospital admission rate, endotracheal intubation rate, mortality and quality of life (COPD-PRO, SF-36).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of moderate to very severe AECOPD
* Age between 40 and 80 years
* Syndrome differentiation meets criteria of syndrome of external cold and internal fluid,syndrome of phlegm-heat congesting lung,or syndrome of phlegm-damp amassing in lung
* Without participations in other interventional trials in the previous one month
* With the informed consent signed

Exclusion Criteria:

* Pregnant and lactating women
* Dementia, mental disorders and reluctant partners
* Complicated with heart failure (NYHA Class IV), or Serious cardiac arrhythmias, or unstable hemodynamics
* Current respiratory disorders other than COPD (e.g., bronchiectasis, active tuberculosis, pneumothorax, Pleural effusion, pulmonary thromboembolic, or Neuromuscular diseases affect respiratory movement function)
* Combined tumor
* Treated outside the hospital for more than 7 days
* Need to carry out invasive mechanical ventilation respiratory failure
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation)
* Bedridden for various reasons
* Allergic to the used medicine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test(CAT) | Change from baseline CAT score at day 0, 14 of the treatment phase, at day 14, 28 of the follow-up phase.
  Using COPD Assessment Test ( CAT) to asses the impact of AECOPD on a person's life, and how this changes over time.

SECONDARY OUTCOMES:
Treatment failure rate | The numbers of treatment failure at day 14 of the treatment phase.
Treatment success rate | The numbers of treatment success at day 14 of the treatment phase.
Length of hospital stays | The length hospital stays in 14 Days of the treatment phase
  length hospital stays will be recorded.
Readmission due to AECOPD | The numbers of readmission due to AECOPD in 28 Days of the followup phase.
  Readmission due to AECOPD will be recorded.
Intubation rate | The numbers of intubation at day 4,7,10，14 of the treatment phase, at day 14, 28 of the follow-up phase.
  Intubation will be recorded.
Mortality | The numbers of mortality at day 14 of the treatment phase and day 28 of the follow-up phase.
Dyspnea | Change from Baseline in the mMRC at day 0, 4, 7, 10,14 of the treatment phase, at day 14, 28 of the follow-up phase.
  Using modified Medical Research Council (mMRC) to asses the dyspnea of COPD, and how this changes over time.
SF-36 | Change from Baseline in the SF-36 at day 0,14 of the treatment phase, at day 14, 28 of the follow-up phase.
  Using the MOS item short from health survey (SF-36) to asses the impact of COPD on a person's life, and how this changes over time.
COPD-PRO | Change from Baseline in the COPD-PRO at day 0,14 of the treatment phase, at day 14, 28 of the follow-up phase.
  Using the COPD patient reported outcome scale (COPD-PRO) to asses the impact of COPD on a person's life, and how this changes over time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Li J, Yu X, Li S, Wang H, Ruan H, Si Y, Xie Y, Wang M. Effects of Chinese medicine on patients with acute exacerbations of COPD: study protocol for a randomized controlled trial. Trials. 2019 Dec 16;20(1):735. doi: 10.1186/s13063-019-3772-y. PMID 31842969